CLINICAL TRIAL: NCT04098354
Title: Telemonitoring and Case Management for Hypertensive and Remote-dwelling Patients With Chronic Kidney Disease - The Telemonitoring for Improved Kidney Outcomes Study (TIKO): A Clinical Research Protocol
Brief Title: Telemonitoring of Hypertensive Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00095231
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This study is designed as a pragmatic randomized controlled trial (RCT) of HBPT plus clinical case management compared to HBPT with usual care. Eligible patients will be randomized 1:1 to HBPT + BP case management versus HBPT + usual care. In the intervention arm, BP will be measured 4 times daily for 1 week, with medications titrated up or down by the study case manager until guideline targets (systolic BP [SBP]: <130mmHg) are achieved. Once BP is controlled, (i.e., to guideline-concordant targets), this 1-week protocol will be repeated every 3 months for 1 year. Patients in the control arm will also follow the same BP measurement protocol, however, there will be no interactions with the case manager; they will share their BP readings with their primary care physicians or nurse practitioners at scheduled visits.
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home-based BP telemonitoring (Active Comparator): Patients will receive a Bluetooth-enabled and validated electronic upper arm oscillometric BP device (A&D Ltd. UA-651BLE; San Jose, CA) that will be paired to their smartphone. Patients will be required to sit with their back rested for at least 5 minutes with the BP cuff around their arm. They will then be required to push the start button on the HBPT device to initiate BP measurement. HBPT values will be based on a series comprised of the mean of duplicate measures, for morning and evening, for a 7-day period and the first day home BP values will not be considered. The BP data will be auto transmitted via Bluetooth to their smartphone and relayed to a secure web portal for review.
  Interventions: Diagnostic Test: home BP telemonitoring system .
- usual care (Placebo Comparator): Patients in the control arm will also follow the same BP measurement protocol as the 'active comparator (intervention) group, however, there will be no interactions with the case manager; they will share their BP readings with their primary care physicians or nurse practitioners at scheduled visits.
  Interventions: Diagnostic Test: home BP telemonitoring system .

INTERVENTIONS:
Diagnostic Test: home BP telemonitoring system . — Patients will receive a Bluetooth-enabled and validated electronic upper arm oscillometric BP device (A&D Ltd. UA-651BLE; San Jose, CA) that will be paired to their smartphone. Patients will be required to sit with their back rested for at least 5 minutes with the BP cuff around their arm. They will then be required to push the start button on the HBPT device to initiate BP measurement. HBPT values will be based on a series comprised of the mean of duplicate measures, for morning and evening, for a 7-day period and the first day home BP values will not be considered. The BP data will be auto transmitted via Bluetooth to their smartphone and relayed to a secure web portal for review.

SUMMARY:
Background:

Hypertension, together with poorly controlled blood pressure (BP) are known risk factors for kidney disease and progression to kidney failure as well as increased cardiovascular (CV) morbidity and mortality. Several studies in patients without kidney disease have demonstrated the efficacy of home BP telemonitoring (HBPT) for BP control.

Objective:

The primary aim of this study is to assess the mean difference in systolic BP (SBP) at 12 months, from baseline in remote dwelling patients with hypertension and chronic kidney disease (CKD) in Northern Alberta, Canada, comparing HBPT + usual care versus HBPT + a case manager. Other secondary objectives, including cost-effectiveness and acceptability of HBPT as well as occurrence of adverse events will also be assessed.

Methods

Design:

This study is designed as a pragmatic randomized controlled trial (RCT) of HBPT plus clinical case management compared to HBPT with usual care.

Setting:

Peace River region in Northern Alberta Region, Canada.

Patients:

Primary care patients with CKD and hypertension.

Measurements:

Eligible patients will be randomized 1:1 to HBPT + BP case management versus HBPT + usual care. In the intervention arm, BP will be measured 4 times daily for 1 week, with medications titrated up or down by the study case manager until guideline targets (systolic BP [SBP]: <130mmHg) are achieved. Once BP is controlled, (i.e., to guideline-concordant targets), this 1-week protocol will be repeated every 3 months for 1 year. Patients in the control arm will also follow the same BP measurement protocol, however, there will be no interactions with the case manager; they will share their BP readings with their primary care physicians or nurse practitioners at scheduled visits.

Limitations:

Potential limitations of this study include the relatively short duration of follow-up, possible technological pitfalls, and need for patients to own a smartphone and have access to the internet to participate.

Conclusions:

As this study will focus on a high-risk population that has been characterized by a large care gap, it will generate important evidence that would allow targeted and effective population-level strategies to be implemented to improve health outcomes for high-risk hypertensive CKD patients in Canada's remote communities.

DETAILED DESCRIPTION:
Introduction:

Poorly controlled blood pressure (BP) is a risk factor for rapid progression of chronic kidney disease (CKD) to kidney failure and is also associated with cardiovascular (CV) morbidity and mortality.Poorly controlled BP is common and often associated with a higher rate of adverse clinical outcomes among remote/rural dwellers due to limited access to and lower quality of chronic disease care. Recent data have demonstrated that remote dwellers with CKD have less access to specialist care, receive poorer clinical care in all aspects of the care process, and exhibit worse clinical outcomes compared to their counterparts living in urban centres. Notably, among remote dwellers with CKD, a lack of BP control is the most important identified element of evidence-based care that is amenable to intervention.

Several studies have demonstrated the feasibility and accuracy of home BP telemonitoring (HBPT) and increased patient satisfaction compared to the usual care among those with some chronic conditions. In one study, when compared to usual care, the adjusted mean SBP differences with HBPT was -4•7 mm Hg [-7•0 to -2•4; P<0.0001] and when HBPT was combined with additional care (e.g. counselling, education, behavioural management, etc) the mean reduction in SBP and DBP was of a larger magnitude, suggesting that HBPT can be more efficacious when proactive additional support is provided. Findings from recent reviews and meta-analyses also show the positive impact of telemonitoring on patient outcomes for those with chronic conditions such as diabetes, asthma, and heart failure. One systematic review and meta-analysis on the effects of HBPT on blood pressure and kidney function in CKD patients reported significant reduction of SBP (-8.8 mmHg; [95% CI: -16.2, -1.4]; P=0.02) and DBP (-2.4 mmHg; [-3.8, -1.0]; P<0.001), and significant improvement in estimated glomerular filtration rate (5.35 mL/min/1.73m2; [2.49, 8.21]; P<0.001). Canadians living in remote communities continue to experience various challenges in accessing healthcare; lack of access to healthcare services and treatments in such settings is often compounded by geographical isolation from mainstream health services. Hence, the use of HBPT technologies could prove to be advantageous for improving control of hypertension and reducing associated target organ damage in populations in remote regions. However, the clinical efficacy, safety, acceptability, and cost-effectiveness of HBPT among CKD patients living in remote/rural communities with limited access to care is unknown.

Therefore, the primary aim of this study is to assess the mean difference in SBP at 12 months, from baseline in remote communities in Northern Alberta through a pragmatic RCT, comparing HBPT + usual care versus HBPT + a case manager.

Methods

Study setting:

This study will be conducted in select remote communities in the Peace River Region of Northern Alberta, located ~1,000 km from Edmonton with a population base of ~75,000. The CKD population in this region receives care from a primary care network consisting of 35 primary care providers (PCPs) affiliated with 9 primary care group practices. Patients with CKD and hypertension will be identified from the Northern Alberta Renal Program (NARP) database and contacted by the study team to participate in this study.

Design, Randomization, and Allocation:

We have designed this study as a two-arm pragmatic RCT comparing the clinical care of remote dwelling hypertensive CKD patients. We will randomly assign the patients with CKD and hypertension to each study arm (1:1) i.e., HBPT plus protocol-based case management versus HBPT plus usual care. A randomized permuted block design of 4 and 6 will be used. The random allocation sequence will be computer generated using STATA 17 software (StataCorp. 2021. Stata Statistical Software: Release 17. College Station, TX: StataCorp LLC) and allocation will be concealed by web-based central randomization using The Research Electronic Data Capture System (REDCap version 8.8.2; 2018 Vanderbilt University).

(i) Intervention arm: Due to the ongoing COVID-19 restrictions for face-to-face patient contact, we will train patients through phone and video contact in addition to sending each participant a written information outlining the study procedures, how to measure their BP, how to download and use the Sphygmo App, and how to transmit BP measurements from their smartphones. Thus, we will train patients to measure BP using guideline recommendations leveraging a locally developed and validated HBPT system (http://mmhg.ca/about-us/). Patients will receive a Bluetooth-enabled and validated electronic upper arm oscillometric BP device (A&D Ltd. UA-651BLE; San Jose, CA) that will be paired to their smartphone. Instructions on how to measure appropriate cuff size will also be provided to each patient. Patients will be required to sit with their back rested for at least 5 minutes with the BP cuff around their arm. They will then be required to push the start button on the HBPT device to initiate BP measurement. HBPT values will be based on a series comprised of the mean of duplicate measures, for morning and evening, for a 7-day period and the first day home BP values will not be considered. Thus, mean SBP for the week will be computed from average of duplicate readings for the next 6 days i.e., 24 measurements. The BP data will be auto transmitted via Bluetooth to their smartphone and relayed to a secure web portal for review. This 7-day protocol will be repeated each month until BP is in the required target range. Once BP is controlled, i.e., guideline-concordant, the 7-day protocol will be repeated every 3 months for 1 year.

Tele-transmitted BP readings will be summarized within the server using telemonitoring software and temporal trends will be plotted. For the active arm of the study, BP data will be tele-transmitted to the study case manager, who will oversee lifestyle modifications and BP self-monitoring and medication adherence. The case manager will also review telemonitored BP summaries, make protocol-based therapeutic adjustments based on a defined algorithm, and send summaries to participants' PCPs to inform them of treatment changes to facilitate communication between patients and care providers. Medications will be adjusted based on guideline recommendations and existing treatment protocols used in other chronic disease settings (i.e., diabetes and stroke). Participants will also receive a document that shows how to unlink their account and delete the Syphmo App from their smartphones at the end of the study.

(ii) Control arm: Patients in the control arm (usual care) will receive the same HBPT device and BP measurement training as those in the intervention arm and will also follow the same measurement protocol. However, the study case manager will not interact with patients in this group. Patients in his group will be expected to inform their PCP or nurse practitioner (NP) of their BP readings at their scheduled consultations. Each participant's PCP / NP will be informed of the patient's involvement in the trial and will receive a letter with a copy of the study synopsis and one-page guideline summary for BP thresholds, targets, and treatments relevant for CKD.

Study procedures and data collection:

At baseline, relevant demographic and health behaviour information including age, sex, race, smoking, alcohol intake and details of patient's medical history and medication history will be collected. Relevant clinical details such as body mass index (BMI) will also be recorded. Blood pressures will be measured and recorded following guideline recommendations. Other information that will be collected includes health care use in the past year (physician and/or emergency room visits, and hospitalizations) ascertained through patient self-reports and/or provincial administrative data sources, quality of life (Kidney Disease Quality of Life-36 [KDQOL-36]) and utility measurements (European Quality of life Five Dimension [EQ-5D]); and satisfaction with receiving health care, using the Patient Assessment of Care for Chronic Conditions (PACIC-2.0).

Laboratory measurements will be carried out at baseline including serum electrolytes, serum creatinine (and estimated glomerular filtration rate), glycated hemoglobin (HbA1c), and urinary albumin/creatinine ratio (UACR). These measurements will also be taken at 6-months and 1 year.

Usability testing will involve assessment of human-computer interaction-specifically, issues related to use, interface, design, function and will also include acceptability of the model of care for the caregivers. We will take a qualitative approach to this process by using focus groups. We plan to recruit two focus groups, one for patients in the telemonitoring arm and one for care providers (case managers and PCPs), with a target sample size of 5 to 8 participants in each group.

Trial-based costing will be assessed with the three-step micro-costing technique of identification, measurement and valuation of relevant health care and non-health care resources using standard methods, with a focus on cost of telemonitoring and case management, health care costs (through linkage with Alberta Health data), and patient-borne costs (patient survey). Thus, the cost-effectiveness (Model A) and cost utility (Model B) of the intervention will be compared against the control using a modified version of a validated economic model used by the team in prior work on HBPT and case management and other chronic diseases. Best practices for economic evaluation will be followed.The intervention includes intermittent or one-time costs (e.g., devices, treatment algorithm development, patient and health care professional training) and ongoing costs (e.g., network and data, case manager time, BP medications). Data captured during the RCT will accurately determine the costs of telemonitoring, case management, and health care use by patients (physician, ER visits, etc.). The change in BP at 1 year, a validated surrogate, will be a key variable in both analyses:

* Model A will calculate the cost per decrement in mean BP using a 1-year time horizon and a public health care payer perspective.
* Model B will estimate incremental cost per quality-adjusted life year (QALY) gained over a lifetime. It will consider longer-term health outcomes, including the probability of developing end-stage kidney disease (ESKD) (requiring dialysis or transplant) or major CV events (i.e., coronary artery disease, heart failure, stroke), all-cause mortality, impacts on quality of life (EQ-5D), and health care costs associated with these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to and more than 18 years with documented diagnosis of established CKD (not on dialysis with eGFR < 60 mL/min/1.73m2 and/or proteinuria > 1 g/day)
* Remote dwelling patients in the Peace River region of Alberta, Canada
* Patients known with hypertension (physician diagnosed / self reported and currently taking antihypertensive medications)
* Owning a smartphone (iOS or Android) with access to wireless internet connection.
* Proficiency in English language (both verbal and written); and ability and willingness to provide informed consent for participation.
* Ability and willingness to use the HBPT device (≥ 80% recordings sent in the training period)

Exclusion Criteria:

* Patients with hypertensive urgency or emergency identified during the training period (immediate consultation will be initiated with the patient's PCP or with a hypertension specialist)
* Patients with stage 5 CKD (eGFR ≤ 15 ml/min/1.73m2) or patients receiving kidney replacement therapy
* Heart failure with reduced ejection fraction
* Presence of any terminal illness (life expectancy < 1 year)
* Participation in any ongoing clinical drug trial
* Pregnancy, lactation / breastfeeding
* Planning to relocate out of the Peace River region or residence in an area without mobile phone coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of telemonitoring and protocol-based case management versus usual care: | Upto 12 months
  The primary outcome will be the mean difference (MD) in home SBP at 12 months, from baseline values.

SECONDARY OUTCOMES:
Proportion of patients with systolic blood pressure within guideline target, user acceptability, adverse events, cost-effectiveness and utility. | upto 12 months
  Secondary outcomes will include (i) proportion of patients with SBP within guideline target at end of the study, from baseline; (ii) Proportion of patients who remained within target SBP throughout the study; (iii) user acceptability of HBPT for BP control; (iv) cost-effectiveness and cost utility of HBPT combined with a protocol-based case management approach, and (v) adverse events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Aminu Bello, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Albert, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okpechi IG, Zaidi D, Ye F, Fradette M, Schick-Makaroff K, Berendonk C, Abdulrahman A, Braam B, Ghimire A, Hariramani VK, Jindal K, Khan M, Klarenbach S, Muneer S, Ringrose J, Scott-Douglas N, Shojai S, Slabu D, Sultana N, Tinwala MM, Thompson S, Padwal R, Bello AK. Telemonitoring and Case Management for Hypertensive and Remote-Dwelling Patients With Chronic Kidney Disease-The Telemonitoring for Improved Kidney Outcomes Study (TIKO): A Clinical Research Protocol. Can J Kidney Health Dis. 2022 Feb 13;9:20543581221077500. doi: 10.1177/20543581221077500. eCollection 2022. PMID 35186305